CLINICAL TRIAL: NCT01939002
Title: An Open-Label, Two-Arm Randomized Study to Characterize Flu-Like Symptoms in Relapsing Multiple Sclerosis Patients Transitioning From Current Interferon Beta Therapies to BIIB017
Brief Title: Characterize Flu-like Symptoms in Relapsing Multiple Sclerosis Patients Transitioning From Non-Pegylated Interferon Beta (IFN-β) Therapies to Peginterferon Beta-1a (BIIB017)
Acronym: ALLOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105MS303
Record Dates: First submitted 2013-08-23; First posted 2013-09-11 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: flu-like symptoms
MeSH Terms: interventions — peginterferon beta-1a; Naproxen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIIB017 plus current FLS therapy (Experimental): Following a 4-week run-in period (starting 1 day after the Screening Visit) in which participants administer non-pegylated IFN therapy, participants receive BIIB017 at an initial dose of 63 μg followed by 94 μg dose at Week 2 and 125 μg every 2 weeks from Week 4 to Week 46, plus current FLS management regimen as determined by the clinician.
  Interventions: Drug: BIIB017
- BIIB017 plus naproxen (Experimental): Following a 4-week run-in period (starting 1 day after the Screening Visit) in which participants administer non-pegylated IFN therapy, participants receive BIIB017 at an initial dose of 63 μg followed by 94 μg dose at Week 2 and 125 μg every 2 weeks from Week 4 to Week 46, plus 500 mg naproxen administered twice daily up to 24 hours prior to BIIB017 treatment and continuing for 48 hours following the BIIB017 injection for the first 8 weeks of treatment, and as recommended by the treating physician subsequently.
  Interventions: Drug: BIIB017; Drug: naproxen

INTERVENTIONS:
Drug: BIIB017
  Other Names: Plegridy; peginterferon beta-1a; PEGylated interferon beta-1a; PEG IFN β-1a
Drug: naproxen
  Other Names: naproxen sodium; Aleve; NSAID; long-acting nonsteroidal anti-inflammatory drug
  Arms: BIIB017 plus naproxen

SUMMARY:
The primary objective of this study is to determine the proportion of participants with relapsing multiple sclerosis who experience new and/or increased flu-like symptoms (FLS) after transitioning from nonpegylated IFN-β therapies to peginterferon beta-1a (BIIB017).

Secondary objectives are: to determine the severity and frequency (measured by flu-like symptom score [FLS-S]) of FLS in these participants; to determine the duration (measured in number of hours) of FLS in these participants; to determine the effect of BIIB017 on other participant-reported outcomes, including treatment satisfaction (measured with the Treatment Satisfaction Questionnaire for Medication [TSQM]) and disability status (measured with the Patient Determined Disease Steps [PDDS]) over a 56-week period; to determine whether interferon-related FLS result in missed days of work/daily activities (e.g., absenteeism); to assess the use of additional medications (in addition to current medications used to treat FLS) to relieve BIIB017-related FLS; to determine the incidence of adverse events throughout the study period; to characterize the immunogenicity profiles of participants switching from prior IFN-β therapy to BIIB017.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a confirmed diagnosis of relapsing forms of multiple sclerosis (MS), as defined by McDonald criteria #1-4 [Polman 2005]
* Must have neurological findings consistent with an Expanded Disability Status Scale (EDSS) score of 0.0 - 5.0
* Must be treated with IFN-β and must be receiving a stable dose of IFN-β for at least 4 months immediately prior to screening
* All male patients and female patients of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 3 months after their last dose of study treatment.

Key Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS [Lublin and Reingold 1996]. These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Patients with these conditions may also have superimposed relapse but are distinguished from patients with relapsing MS by the lack of clinically stable periods or clinical improvement
* History of severe allergic or anaphylactic reactions or known hypersensitivity to medication which might suggest potential for a reaction to IFN β-1a or polyethylene glycol
* History of malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured)
* History of seizure disorder or unexplained blackouts OR history of a seizure within 3 months prior to Baseline
* Known allergy to any component of the BIIB017 formulation
* An MS relapse that has occurred within the 50 days prior to Baseline (Day 1) and/or lack of stabilization from a previous relapse prior to Baseline.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (37):
- United States (37):
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Boulder, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Dover, Delaware
  - Research Site, Newark, Delaware
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Chesterfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Latham, New York
  - Research Site, Plainview, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Greenville, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Newport News, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 251 participants who entered into the run-in period of non-pegylated interferon (IFN) therapy, a total of 201 were randomized.
Groups:
- BIIB017 Plus Current FLS Therapy: Following a 4-week run-in period (starting 1 day after the Screening Visit) in which participants administered non-pegylated IFN therapy, participants received BIIB017 at an initial dose of 63 μg followed by 94 μg dose at Week 2 and 125 μg every 2 weeks from Week 4 to Week 46, plus current FLS management regimen as determined by the clinician.
- BIIB017 Plus Naproxen: Following a 4-week run-in period (starting 1 day after the Screening Visit) in which participants administered non-pegylated IFN therapy, participants received BIIB017 at an initial dose of 63 μg followed by 94 μg dose at Week 2 and 125 μg every 2 weeks from Week 4 to Week 46, plus 500 mg naproxen administered twice daily up to 24 hours prior to BIIB017 treatment and continuing for 48 hours following the BIIB017 injection for the first 8 weeks of treatment, and as recommended by the treating physician subsequently.
Period: Overall Study
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Started | 103 | 98
Completed | 84 | 80
Not Completed | 19 | 18
Not completed — Adverse Event | 13 | 13
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Total
Number analyzed (Participants) | 103 | 98 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.76 (10.32) | 49.88 (9.45) | 49.82 (9.88)
Gender [Count of Participants; unit: Participants]
  Female | 84 | 79 | 163
  Male | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing New or Increased FLS During the First 8 Weeks: Overall Population
Description: The total Flu-like Symptoms Score (FLS-S) is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. New or increased FLS is defined as an FLS overall score of 2 points or greater over Screening. Pre-dose data were not used; up to 48-hour data after dosing were used. Overall score was imputed as the average score after dose.
Time Frame: during the first 8 weeks of treatment
Population: Efficacy population: randomized participants who received at least 1 dose of study treatment and had efficacy data in both the 4-week run-in period and the post-baseline treatment period.
Measure: Number; unit: percentage of participants
Groups:
- Overall Population: Following a 4-week run-in period (starting 1 day after the Screening Visit) in which participants administered non-pegylated IFN therapy, participants received BIIB017 at an initial dose of 63 μg followed by 94 μg dose at Week 2 and 125 μg every 2 weeks from Week 4 to Week 46, plus:
  * current FLS management regimen as determined by the clinician; or
  * 500 mg naproxen administered twice daily up to 24 hours prior to BIIB017 treatment and continuing for 48 hours following the BIIB017 injection for the first 8 weeks of treatment, and as recommended by the treating physician subsequently.
Arm/Group | Overall Population
Number analyzed (Participants) | 194
percentage of participants | 10.3
Statistical Analysis 1: Comparison: Overall Population; Test type: Superiority or Other; p < 0.0001, Chi-squared — 1-sample Chi-square test comparing to Null hypotheses at 25%

2. Secondary Outcome: Percentage of Participants Experiencing New or Increased FLS During the First 8 Weeks: Between FLS Management Arms
Description: The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. New or increased FLS is defined as an FLS overall score of 2 points or greater over Screening. Pre-dose data were not used; up to 48-hour data after dosing were used. Overall score was imputed as the average score after dose.
Time Frame: during the first 8 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
percentage of participants | 13 | 7.4
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.2037, Chi-squared — Chi-square test between 2 treatment arms

3. Secondary Outcome: Percentage of Participants With Any FLS in the 4-Week Run-In Period, During the First 8 Weeks of Treatment, and During 48 Weeks of Treatment
Description: Any FLS is defined as an FLS-S total score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. 4WRI=4-week run-in; F8W=first 8 weeks; 48W=48 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment, 48 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
percentage of participants
  4WRI | 88 | 91.5 | 89.7
  F8W | 91 | 88.3 | 89.7
  48W | 95 | 94.7 | 94.8

4. Secondary Outcome: Shift in Percentage of Participants With Any FLS From 4-Week Run-In Period to the First 8 Weeks
Description: Any FLS is defined as an FLS-S total score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. Pre-dose data not were used. Data up to 48-hours after dosing were used. Total score was imputed as the highest score after dose. 4WRI=4-week run-in period; F8W=first 8 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
percentage of participants
  With FLS in 4WRI / With FLS during F8W | 85.00 | 82.98 | 84.02
  With FLS in 4WRI / Without FLS during F8W | 3.00 | 8.51 | 5.67
  Without FLS in 4WRI / With FLS during F8W | 6.00 | 5.32 | 5.67
  Without FLS in 4WRI / Without FLS during F8W | 6.00 | 3.19 | 4.64
Statistical Analysis 1: Comparison: Overall Population; Test type: Superiority or Other; p = 1.00, McNemar; McNemar tests the null hypothesis of no difference in FLS between 4WRI and F8W
Statistical Analysis 2: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.5078, McNemar
Statistical Analysis 3: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.5811, McNemar

5. Secondary Outcome: Shift in Percentage of Participants With Any FLS From 4-Week Run-In Period to 48 Weeks
Description: Any FLS is defined as an FLS-S total score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. Pre-dose data not were used. Data up to 48-hours after dosing were used. Total score was imputed as the highest score after dose. 4WRI=4-week run-in period; 48W=48 weeks.
Time Frame: 4-week run-in period, 48 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
percentage of participants
  With FLS in 4WRI / With FLS during 48W | 86.00 | 87.23 | 86.60
  With FLS in 4WRI / Without FLS during 48W | 2.00 | 4.26 | 3.09
  Without FLS in 4WRI / With FLS during 48W | 9.00 | 7.45 | 8.25
  Without FLS in 4WRI / Without FLS during 48W | 3.00 | 1.06 | 2.06
Statistical Analysis 1: Comparison: Overall Population; Test type: Superiority or Other; p = 0.0525, McNemar
Statistical Analysis 2: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0654, McNemar
Statistical Analysis 3: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.5488, McNemar

6. Secondary Outcome: Summary of Severity of FLS (Per FLS-S) in the First 8 Weeks Compared to 4-Week Run-In Period Between Arms
Description: The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. 4WRI=4-week run-in period; F8W=first 8 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Severity of FLS in 4WRI | 1.198 (1.224) | 1.05 (1.02) | 1.126 (1.129)
  Severity of FLS in F8W | 1.311 (1.185) | 1.036 (0.951) | 1.178 (1.084)
  Mean Change from 4WRI to F8W | 0.113 (0.67) | -0.013 (0.581) | 0.052 (0.63)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0945, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.8246, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.2533, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.1631, 2-sample t-test between 2 arms

7. Secondary Outcome: Summary of Severity of FLS (Per FLS-S) in the 48 Weeks of Treatment Compared to 4-Week Run-In Period Between Arms
Description: The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. 4WRI=4-week run-in period; 48W=48 weeks.
Time Frame: 4-week run-in period, 48 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Severity of FLS in 4WRI | 1.2 (1.22) | 1.05 (1.02) | 1.13 (1.13)
  Severity of FLS in 48W | 1.28 (1.19) | 0.98 (1.00) | 1.14 (1.11)
  Mean Change from 4WRI to 48W | 0.08 (0.83) | -0.07 (0.7) | 0.01 (0.77)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.3189, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.3582, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.8484, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.1771, 2-sample t-test between 2 arms

8. Secondary Outcome: Summary of Average Duration of FLS in the First 8 Weeks of Treatment
Description: Duration of FLS for a treatment was defined as the sum of hours from the time of treatment to 48 hours with an FLS-S score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. If an FLS is > 0 at an evaluation time, 6 hours were counted as the duration assuming the event started from previous evaluation time. Average duration of FLS for the first 8 weeks was defined as the mean duration from Weeks 0, 2, 4, 6, and 8. 4WRI=4-week run-in period; F8W=first 8 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment
Population: Efficacy population: randomized participants who received at least 1 dose of study treatment and had efficacy data in both the 4-week run-in period and the post-baseline treatment period; n=number of subjects assessed at the given timepoint.
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
hours
  Average duration in 4WRI; n=88, 86, 174 | 16 [6 to 33.38] | 12.8 [6 to 42.86] | 13.75 [6 to 42.86]
  Average duration in F8W; n=91, 83, 174 | 18 [6 to 40.8] | 18 [6 to 43.5] | 18 [6 to 43.5]
  Change from 4WRI to F8W; n=85, 78, 163 | 2.1 [-16.5 to 18.4] | 3.8 [-10.5 to 20.4] | 3 [-16.5 to 20.4]
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0009, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.3792, 2-sample t-test between 2 arms

9. Secondary Outcome: Summary of Average Duration of FLS in the 48 Weeks of Treatment
Description: Duration of FLS for a treatment was defined as the sum of hours from the time of treatment to 48 hours with a FLS-S score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. If a FLS is > 0 at an evaluation time, 6 hours were counted as the duration assuming the event started from previous evaluation time. Average duration of FLS for the first 8 weeks was defined as the mean duration from Weeks 0, 2, 4, 6, and 8. 4WRI=4-week run-in period; 48W=48 weeks.
Time Frame: 4-week run-in period, 48 weeks of treatment
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
hours
  Average duration in 4WRI; n=88, 86, 174 | 16 [6 to 33.38] | 12.8 [6 to 42.86] | 13.75 [6 to 42.86]
  Average duration in 48W; n=95, 89, 184 | 16.75 [6 to 38.09] | 16.96 [6 to 39] | 16.96 [6 to 39]
  Change from 4WRI to 48W; n=86, 82, 168 | 2.82 [-19.57 to 17.83] | 2 [-10 to 14.88] | 2.16 [-19.57 to 17.83]
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0019, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.0009, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm

10. Secondary Outcome: Summary of FLS-Visual Analogue Scale (VAS) During the First 8 Weeks of Treatment Compared to 4-Week Run-In Period: Effectiveness of FLS Treatment
Description: Participants reported the effectiveness of their FLS management regimen on a 100-mm VAS between not effective (0) and very effective (100). 4WRI=4-week run-in period; F8W=first 8 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment
Population: Efficacy population: randomized participants who received at least 1 dose of study treatment and had efficacy data in both the 4-week run-in period and the post-baseline treatment period; n=number of participants assessed at the given timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Effectiveness in 4WRI; n=91, 86, 177 | 64.5 (27.952) | 66.398 (28.855) | 65.422 (28.329)
  Effectiveness in F8W; n=96, 91, 187 | 69.695 (22.423) | 74.253 (23.85) | 71.913 (23.179)
  Change from 4WRI to F8W; n=87, 83, 170 | 6.525 (23.271) | 5.694 (29.151) | 6.119 (26.231)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0105, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.0789, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.0027, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.8380, 2-sample t-test between 2 arms

11. Secondary Outcome: Summary of FLS-VAS During the First 8 Weeks of Treatment Compared to 4-Week Run-In Period: Satisfaction With FLS Treatment
Description: Participants reported their satisfaction with the effectiveness of their FLS management regimen on a 100-mm VAS between not satisfied (0) and very satisfied (100). 4WRI=4-week run-in period; F8W=first 8 weeks.
Time Frame: 4-week run-in period, first 8 weeks of treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Satisfaction in 4WRI; n=91, 86, 177 | 68.654 (26.574) | 72.778 (23.817) | 70.658 (25.285)
  Satisfaction in F8W; n=96, 91, 187 | 71.153 (21.884) | 74.684 (23.671) | 72.871 (22.778)
  Change from 4WRI to F8W; n=87, 83, 170 | 3.715 (23.307) | 0.759 (24.729) | 2.272 (23.986)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.1407, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.7805, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.2186, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.4234, 2-sample t-test between 2 arms

12. Secondary Outcome: Summary of FLS-VAS During the 48 Weeks of Treatment Compared to 4-Week Run-In Period: Effectiveness of FLS Treatment
Description: Participants reported the effectiveness of their FLS management regimen on a 100-mm VAS between not effective (0) and very effective (100). 4WRI=4-week run-in period; 48W=48 weeks.
Time Frame: 4-week run-in period, 48 weeks of treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Effectiveness in 4WRI; n=91, 86, 177 | 64.5 (27.952) | 66.398 (28.855) | 65.422 (28.329)
  Effectiveness in 48W; n=99, 94, 193 | 70.547 (21.657) | 75.416 (21.28) | 72.918 (21.557)
  Change from 4WRI to 48W; n=90, 86, 176 | 6.803 (24.182) | 8.042 (27.206) | 7.408 (25.638)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0090, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.0075, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.0002, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.7497, 2-sample t-test between 2 arms

13. Secondary Outcome: Summary of FLS-VAS During the 48 Weeks of Treatment Compared to 4-Week Run-In Period: Satisfaction With FLS Treatment
Description: Participants reported their satisfaction with the effectiveness of their FLS management regimen on a 100-mm VAS between not satisfied (0) and very satisfied (100). 4WRI=4-week run-in period; 48W=48 weeks.
Time Frame: 4-week run-in period, 48 weeks of treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 100 | 94 | 194
units on a scale
  Satisfaction in 4WRI; n=91, 86, 177 | 68.654 (26.574) | 72.778 (23.817) | 70.658 (25.285)
  Satisfaction in 48W; n=99, 94, 193 | 72.192 (21.053) | 76.061 (21.075) | 74.076 (21.098)
  Change from 4WRI to 48W; n=90, 86, 176 | 4.607 (22.43) | 2.274 (21.874) | 3.467 (22.128)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Test type: Superiority or Other; p = 0.0545, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.3377, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Test type: Superiority or Other; p = 0.0391, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Test type: Superiority or Other; p = 0.4861, 2-sample t-test between 2 arms

14. Secondary Outcome: Percentage of Participants Requiring Additional FLS Management Regimen to Relieve BIIB017-related FLS
Time Frame: during the first 8 weeks of treatment
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
percentage of participants
  Used additional regimen, first 8 weeks; n=78, 85 | 6.4 | 15.3
  No additional regimen, first 8 weeks; n=78, 85 | 93.6 | 84.7
  Used additional regimen, Weeks 0-2; n=57, 73 | 1.8 | 11
  No additional regimen, Weeks 0-2; n=57, 73 | 98.2 | 89
  Used additional regimen, Weeks 3-4; n=61, 77 | 6.6 | 5.2
  No additional regimen, Weeks 3-4; n=61, 77 | 93.4 | 94.8
  Used additional regimen, Weeks 5-6; n=63, 76 | 0 | 2.6
  No additional regimen, Weeks 5-6; n=63, 76 | 100 | 97.4
  Used additional regimen, Weeks 7-8; n=52, 74 | 1.9 | 4.1
  No additional regimen, Weeks 7-8; n=52, 74 | 98.1 | 95.9
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; first 8 weeks; Test type: Superiority or Other; p = 0.0834, Fisher Exact
Statistical Analysis 2: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Weeks 0-2; Test type: Superiority or Other; p = 0.0767, Fisher Exact
Statistical Analysis 3: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Weeks 3-4; Test type: Superiority or Other; p = 0.7320, Fisher Exact
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Weeks 5-6; Test type: Superiority or Other; p = 0.5008, Fisher Exact
Statistical Analysis 5: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Weeks 7-8; Test type: Superiority or Other; p = 0.6422, Fisher Exact

15. Secondary Outcome: Mean Change From 4-Week Run-In Period at Each Visit for Treatment Satisfaction Questionnaire for Medication (TSQM), Effectiveness Scale Factor: Overall Population
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to each visit using transformed scores between 0 and 100 for effectiveness (with higher scores indicating greater satisfaction) are presented. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Weeks 4, 12, 24, 36, 48 (or Early Termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 194
units on a scale
  Effectiveness at 4WRI; n=194 | 73.871 (20.131)
  Change at Week 4; n=185 | -2.589 (28.139)
  Change at Week 12; n=175 | -1.274 (30.682)
  Change at Week 24; n=167 | 0.341 (27.401)
  Change at Week 36; n =162 | 1.864 (29.175)
  Change at Week 48; n=153 | 2.863 (29.172)
  Change at Early Termination; n=26 | -17.308 (34.534)
Statistical Analysis 1: Comparison: Overall Population; change at Week 4; Test type: Superiority or Other; p = 0.2123, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.5834, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p = 0.8723, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p = 0.4173, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.2267, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; change at Early Term; Test type: Superiority or Other; p = 0.0171, paired t-test within 1 arm

16. Secondary Outcome: Mean Change From 4-Week Run-In Period at Each Visit for TSQM, Side-Effects Scale Factor: Overall Population
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to each visit using transformed scores between 0 and 100 for side effects (with higher scores indicating greater satisfaction) are presented. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Weeks 4, 12, 24, 36, 48 (or Early Termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 194
units on a scale
  Side Effects at 4WRI; n=194 | 85.17 (18.136)
  Change at Week 4; n=185 | 6.065 (21.243)
  Change at Week 12; n=175 | 5.109 (19.67)
  Change at Week 24; n=167 | 2.958 (18.131)
  Change at Week 36; n=162 | 3.37 (18.207)
  Change at Week 48; n=153 | 1.418 (20.922)
  Change at Early Termination; n=26 | -18.731 (31.776)
Statistical Analysis 1: Comparison: Overall Population; change at Week 4; Test type: Superiority or Other; p = 0.0001, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.0007, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p = 0.0365, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p = 0.0197, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.4031, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p = 0.0060, paired t-test within 1 arm

17. Secondary Outcome: Mean Change From 4-Week Run-In Period at Each Visit for TSQM, Convenience Scale Factor: Overall Population
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to each visit using transformed scores between 0 and 100 for convenience (with higher scores indicating greater satisfaction) are presented. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Weeks 4, 12, 24, 36, 48 (or Early Termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 194
units on a scale
  Convenience at 4WRI; n=194 | 66.665 (16.588)
  Change at Week 4; n=185 | 18.703 (21.864)
  Change at Week 12; n=175 | 18.12 (20.588)
  Change at Week 24; n=167 | 18.419 (20.804)
  Change at Week 36; n =162 | 18.704 (21.258)
  Change at Week 48; n=153 | 19.588 (20.912)
  Change at Early Termination; n=26 | 7.808 (28.788)
Statistical Analysis 1: Comparison: Overall Population; change at Week 4; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p = 0.1789, paired t-test within 1 arm
Statistical Analysis 7: Comparison: Overall Population; Test type: Superiority or Other; p = 0.2248, general linear model — p-value on slope is based on general linear model with repeat measures over all visits

18. Secondary Outcome: Mean Change From 4-Week Run-In Period at Each Visit for TSQM, Global Satisfaction Scale Factor: Overall Population
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to each visit using transformed scores between 0 and 100 for global satisfaction (with higher scores indicating greater satisfaction) are presented. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Weeks 4, 12, 24, 36, 48 (or Early Termination)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 194
units on a scale
  Global Satisfaction at 4WRI; n=194 | 75.985 (15.137)
  Change at Week 4; n=185 | 6.789 (19.8)
  Change at Week 12; n=175 | 7.354 (20.296)
  Change at Week 24; n=167 | 7.575 (19.91)
  Change at Week 36; n =162 | 9.179 (19.215)
  Change at Week 48; n=153 | 8.556 (23.389)
  Change at Early Termination; n=26 | -38.538 (26.224)
Statistical Analysis 1: Comparison: Overall Population; change at Week 4; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 7: Comparison: Overall Population; Test type: Superiority or Other; p < 0.0001, general linear model — p-value on slope is based on general linear model with repeat measures over all visits

19. Secondary Outcome: Mean Change From 4-Week Run-In Period at Week 4 for TSQM, Effectiveness Scale Factor: Between FLS Management Arms
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to Week 4 using transformed scores between 0 and 100 for effectiveness (with higher scores indicating greater satisfaction) are presented. This secondary endpoint was targeted for Week 4 only. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
units on a scale
  Effectiveness at 4WRI; n=100, 94 | 75.16 (19.431) | 72.5 (20.866)
  Change at Week 4; n=95, 90 | 0.979 (24.793) | -6.356 (30.982)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; change at Week 4; Test type: Superiority or Other; p = 0.7012, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.0548, paired t-test within 1 arm
Statistical Analysis 3: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.0782, 2-sample t-test between 2 arms

20. Secondary Outcome: Mean Change From 4-Week Run-In Period at Week 4 for TSQM, Side Effects Scale Factor: Between FLS Management Arms
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to Week 4 using transformed scores between 0 and 100 for side effects (with higher scores indicating greater satisfaction) are presented. This secondary endpoint was targeted for Week 4 only. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
units on a scale
  Side Effects at 4WRI; n=100, 94 | 83.78 (20.074) | 86.649 (15.789)
  Change at Week 4; n=95, 90 | 8.579 (23.576) | 3.411 (18.222)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; change at Week 4; Test type: Superiority or Other; p = 0.0006, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.0792, paired t-test within 1 arm
Statistical Analysis 3: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.0961, 2-sample t-test between 2 arms

21. Secondary Outcome: Mean Change From 4-Week Run-In Period at Week 4 for TSQM, Convenience Scale Factor: Between FLS Management Arms
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to Week 4 using transformed scores between 0 and 100 for convenience (with higher scores indicating greater satisfaction) are presented. This secondary endpoint was targeted for Week 4 only. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
units on a scale
  Convenience at 4WRI; n=100, 94 | 65.94 (15.878) | 67.436 (17.365)
  Change at Week 4; n=95, 90 | 19.768 (22.403) | 17.578 (21.347)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; change at Week 4; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 3: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.4973, 2-sample t-test between 2 arms

22. Secondary Outcome: Mean Change From 4-Week Run-In Period at Week 4 for TSQM, Global Satisfaction Scale Factor: Between FLS Management Arms
Description: The TSQM assessed participants' global satisfaction with treatment and captured information on treatment side effects, effectiveness, and convenience. Changes from the 4-week run-in period to Week 4 using transformed scores between 0 and 100 for global satisfaction (with higher scores indicating greater satisfaction) are presented. This secondary endpoint was targeted for Week 4 only. 4WRI=4-week run-in.
Time Frame: 4-week run-in period, Week 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 100 | 94
units on a scale
  Global Satisfaction at 4WRI; n=100, 94 | 75.86 (14.001) | 76.117 (16.334)
  Change at Week 4; n=95, 90 | 8.663 (16.633) | 4.811 (22.596)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; change at Week 4; Test type: Superiority or Other; p < 0.0001, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.0464, paired t-test within 1 arm
Statistical Analysis 3: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; change at Week 4; Test type: Superiority or Other; p = 0.1905, 2-sample t-test between 2 arms

23. Secondary Outcome: Mean Change From Screening at Each Visit in Absenteeism Questionnaire, Usual Work Days Per Week: Overall Population
Description: Categorical questions in the Absenteeism Questionnaire asked participants to report the number of usual work days per week, the number of days missed in 2 weeks from multiple sclerosis (MS) symptoms, and the number of days missed in 2 weeks from MS treatment. This secondary endpoint was targeted to analyze the Overall Population only. 4WRI=4-week run-in.
Time Frame: Week -4 (screening), Week 12, Week 24, Week 36, Week 48, Early Termination
Population: Efficacy population: randomized participants who received at least 1 dose of study treatment, had efficacy data in both the 4-week run-in period and the post-baseline treatment period, and were employed; n=number of participants assessed at the given timepoint.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Overall Population
Number analyzed (Participants) | 123
days
  Days in 4WRI; n=123 | 4.691 (1.033)
  Change at Week 12; n=106 | -0.019 (0.436)
  Change at Week 24; n=99 | -0.081 (0.566)
  Change at Week 36; n=96 | -0.052 (0.773)
  Change at Week 48; n=95 | 0.032 (0.573)
  Change at Early Termination; n=15 | 0.2 (0.862)
Statistical Analysis 1: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.6569, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p = 0.1584, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p = 0.5106, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.5927, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p = 0.3840, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; Test type: Superiority or Other; p = 0.4182, general linear model — p-value on slope is based on general linear model with repeat measures over all visits

24. Secondary Outcome: Mean Change From Screening at Each Visit in Absenteeism Questionnaire, Days Missed in 2 Weeks From MS Symptoms: Overall Population
Description: Categorical questions in the Absenteeism Questionnaire asked participants to report the number of usual work days per week, the number of days missed in 2 weeks from MS symptoms, and the number of days missed in 2 weeks from MS treatment. This secondary endpoint was targeted to analyze the Overall Population only. 4WRI=4-week run-in.
Time Frame: Week -4 (screening), Week 12, Week 24, Week 36, Week 48, Early Termination
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Overall Population
Number analyzed (Participants) | 123
days
  Days in 4WRI; n=123 | 0.016 (0.127)
  Change at Week 12; n=106 | 0.057 (0.513)
  Change at Week 24; n=99 | 0.061 (0.373)
  Change at Week 36; n=96 | 0 (0.205)
  Change at Week 48; n =95 | 0.137 (1.078)
  Change at Early Termination; n=15 | 0 (0)
Statistical Analysis 1: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.2588, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p = 0.1092, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p = 1.0000, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.2190, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; Test type: Superiority or Other; p = 0.6402, general linear model — p-value on slope is based on general linear model with repeat measures over all visits

25. Secondary Outcome: Mean Change From Screening at Each Visit in Absenteeism Questionnaire, Days Missed in 2 Weeks From MS Treatment: Overall Population
Description: as for outcome 24
Time Frame: Week -4 (screening), Week 12, Week 24, Week 36, Week 48, Early Termination
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Overall Population
Number analyzed (Participants) | 123
days
  Days in 4WRI; n=123 | 0.016 (0.127)
  Change at Week 12; n=106 | 0.019 (0.275)
  Change at Week 24; n=99 | 0.02 (0.319)
  Change at Week 36; n=96 | -0.021 (0.144)
  Change at Week 48; n =95 | 0.126 (1.074)
  Change at Early Termination; n=15 | 0.2 (0.414)
Statistical Analysis 1: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.4821, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 24; Test type: Superiority or Other; p = 0.5298, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Week 36; Test type: Superiority or Other; p = 0.1584, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.2547, paired t-test within 1 arm
Statistical Analysis 5: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p = 0.0824, paired t-test within 1 arm
Statistical Analysis 6: Comparison: Overall Population; Test type: Superiority or Other; p = 0.3148, general linear model — p-value on slope is based GLM with repeat measures over all visits

26. Secondary Outcome: Change From Baseline Visit (Day 1) to Week 48 in Walking Disability Status as Measured by Patient Determined Disease Steps (PDDS): Overall Population
Description: Subjects rated their perceived walking disability on a scale of 0 to 8 using the PDDS, with higher scores indicating more severe disability. This secondary endpoint was targeted to analyze the Overall Population only.
Time Frame: Day 1 (Baseline, pre-dose), Week 12, Week 48, Early Termination
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 194
units on a scale
  Baseline; n=194 | 0.83 (1.258)
  Change at Week 12; n=174 | 0.029 (0.836)
  Change at Week 48; n=153 | 0.15 (0.857)
  Change Early Termination; n=26 | 0.346 (1.093)
Statistical Analysis 1: Comparison: Overall Population; change at Week 12; Test type: Superiority or Other; p = 0.6508, paired t-test within 1 arm
Statistical Analysis 2: Comparison: Overall Population; change at Week 48; Test type: Superiority or Other; p = 0.0315, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; change at Early Termination; Test type: Superiority or Other; p = 0.1190, paired t-test within 1 arm
Statistical Analysis 4: Comparison: Overall Population; Test type: Superiority or Other; p = 0.1520, general linear model — p-value on slope is based GLM with repeat measures over all visits

27. Secondary Outcome: Summary of Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations Due to AEs
Description: An AE was any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, placed the subject at immediate risk of death (a life-threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, could jeopardize the subject or could require intervention to prevent one of the other outcomes listed in the definition above. ISR=injection site reactions.
Time Frame: Day 1 to Week 52
Population: Safety population: all participants who received at least 1 injection of study treatment.
Measure: Number; unit: participants
Groups:
- BIIB017 Plus Current FLS Therapy: BIIB017 initial dose of 63 μg followed by 94 μg dose at week 2 and 125 μg every 2 weeks from week 4 to week 46, plus current FLS management regimen as determined by the clinician
- BIIB017 Plus Naproxen: BIIB017 initial dose of 63 μg followed by 94 μg dose at week 2 and 125 μg every 2 weeks from week 4 to week 46, plus 500 mg naproxen administered twice daily up to 24 hours prior to BIIB017 treatment and continuing for 48 hours following the BIIB017 injection for the first 8 weeks of treatment, and as recommended by the treating physician subsequently
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Number analyzed (Participants) | 103 | 98
participants
  Any event | 93 | 90
  Moderate or severe event | 54 | 60
  Severe event | 7 | 12
  Related event | 80 | 71
  Serious event | 4 | 6
  Discontinuations due to AEs | 14 | 13
  Treatment discontinuation due to FLS event | 3 | 2
  Treatment discontinuation due to ISR events | 5 | 3
  Study discontinuation due to an event | 13 | 13

28. Secondary Outcome: Summary of Average Duration of FLS Within the Last 4 Weeks of the BIIB017 Treatment Period Compared With the Duration of FLS in the 4-Week Run-In Period
Description: Average duration of FLS for the last 4 weeks (L4W) is defined as the mean duration of last 4 weeks. Duration of FLS for a treatment is defined as the sum of hours from the treatment to 48 hours with a FLS-S score > 0. The total FLS-S is the sum of all 4 symptom scores (muscle aches, chills, fatigue and fever), each rated from 0 (absent) to 3 (severe), with a range of 0-12 with 0 indicating no FLS and 12 indicating severe FLS. If a FLS is > 0 at an evaluation time, 6 hours were counted as the duration assuming the event started from previous evaluation time. 4WRI=4-week run-in.
Time Frame: Weeks -4 to -1 (Screening), Weeks 45-48 (last 4 weeks of study)
Population: Efficacy population: randomized participants who received at least 1 dose of study treatment, had efficacy data in both the 4-week run-in period and the post-baseline treatment period, and had FLS; n=number of participants assessed at the given timepoint.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen | Overall Population
Number analyzed (Participants) | 88 | 86 | 174
hours
  Average duration in 4WRI; n=88, 86, 174 | 16.067 (8.277) | 14.915 (7.637) | 15.497 (7.965)
  Average duration in L4W; n=87, 83, 170 | 18.057 (9.06) | 15.892 (8.073) | 17 (8.635)
  Change from 4WRI to L4W; n=80, 77, 157 | 2.612 (8.067) | 0.943 (6.738) | 1.793 (7.468)
Statistical Analysis 1: Comparison: BIIB017 Plus Current FLS Therapy; Change from 4WRI to L4W; Test type: Superiority or Other; p = 0.0049, paired t-test within 1 arm
Statistical Analysis 2: Comparison: BIIB017 Plus Naproxen; Change from 4WRI to L4W; Test type: Superiority or Other; p = 0.2230, paired t-test within 1 arm
Statistical Analysis 3: Comparison: Overall Population; Change from 4WRI to L4W; Test type: Superiority or Other; p = 0.0031, paired t-test within 1 arm
Statistical Analysis 4: Comparison: BIIB017 Plus Current FLS Therapy vs BIIB017 Plus Naproxen; Change from 4WRI to L4W; Test type: Superiority or Other; p = 0.1624, 2-sample t-test between 2 arms

29. Secondary Outcome: Antibody Data in the Overall Population: IFN β-1a Antibody Screening
Description: The number of participants who tested positive for IFN β-1a binding antibodies (BAbs). Value was coded as 'positive' if observed value > 0 or coded as 'negative' if observed value < 0. This secondary endpoint was targeted to analyze the Overall Population only.
Time Frame: Baseline (BL; Day 1), Week 12, Week 24, Week 36, Week 48 or early withdrawal (EW)
Population: Safety population: participants who received at least 1 injection of study treatment and had an assessment; n=number of participants with an assessment at given timepoint.
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 199
participants
  Baseline: Positive; n=199 | 22
  Baseline: Negative; n=199 | 177
  Any post-baseline visit: Positive; n=198 | 35
  Any post-baseline visit: Negative; n=198 | 178
  Week 12: Positive; n=183 | 26
  Week 12: Negative; n=183 | 157
  Week 24: Positive; n=171 | 22
  Week 24: Negative; n=171 | 149
  Week 36: Positive; n=167 | 18
  Week 36: Negative; n=167 | 149
  Week 48/EW: Positive; n=193 | 25
  Week 48/EW: Negative; n=193 | 168
  Negative at BL with ≥ 1 positive post-BL; n=174 | 13

30. Secondary Outcome: Antibody Data in the Overall Population: IFN β-1a Anti-Pegylated (PEG) Antibody Testing
Description: The number of participants who tested positive or negative for IFN β-1a anti-PEG antibodies. Value was coded as 'positive' if observed value > 0 or coded as 'negative' if observed value < 0. This secondary endpoint was targeted to analyze the Overall Population only.
Time Frame: Baseline (BL; Day 1), Week 12, Week 24, Week 36, Week 48 or early withdrawal (EW)
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 201
participants
  Baseline: Positive; n=201 | 7
  Baseline: Negative; n=201 | 194
  Any post-baseline visit: Positive; n=198 | 8
  Any post-baseline visit: Negative; n=198 | 196
  Week 12: Positive; n=182 | 6
  Week 12: Negative; n=182 | 176
  Week 24: Positive; n=173 | 3
  Week 24: Negative; n=173 | 170
  Week 36: Positive; n=168 | 1
  Week 36: Negative; n=168 | 167
  Week 48/EW: Positive; n=193 | 3
  Week 48/EW: Negative; n=193 | 190
  Negative at BL with ≥ 1 positive post-BL; n=192 | 4

31. Secondary Outcome: Antibody Data in the Overall Population: IFN β-1a Neutralizing Antibodies (Nabs) Testing
Description: The number of participants who tested positive for IFN β-1a Nabs. Value was coded as 'positive' if observed value > 0 or coded as 'negative' if observed value < 0. This secondary endpoint was targeted to analyze the Overall Population only.
Time Frame: Baseline (Day 1), Week 12, Week 24, Week 36, Week 48 or early withdrawal (EW)
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Overall Population
Number analyzed (Participants) | 201
participants
  Baseline: Positive; n=22 | 14
  Baseline: Negative; n=22 | 8
  Any post-baseline visit: Positive; n=35 | 17
  Any post-baseline visit: Negative; n=35 | 20
  Week 12: Positive; n=26 | 15
  Week 12: Negative; n=26 | 11
  Week 24: Positive; n=22 | 11
  Week 24: Negative; n=22 | 11
  Week 36: Positive; n=18 | 11
  Week 36: Negative; n=18 | 7
  Week 48/EW: Positive; n=25 | 12
  Week 48/EW: Negative; n=25 | 13
  Negative at BL with ≥ 1 positive post-BL; n=7 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Week 52
Arm/Group | BIIB017 Plus Current FLS Therapy | BIIB017 Plus Naproxen
Serious Adverse Events (participants affected / at risk) | 4/103 | 6/98
Other Adverse Events (participants affected / at risk) | 92/103 | 90/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB017 Plus Current FLS Therapy (N=103) | BIIB017 Plus Naproxen (N=98)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIIB017 Plus Current FLS Therapy (N=103) | BIIB017 Plus Naproxen (N=98)
Injection site erythema (General disorders) | 46 | 34
Injection site reaction (General disorders) | 23 | 21
Influenza like illness (General disorders) | 11 | 13
Injection site pruritus (General disorders) | 12 | 7
Injection site pain (General disorders) | 8 | 3
Injection site bruising (General disorders) | 4 | 6
Fatigue (General disorders) | 2 | 6
Pain (General disorders) | 2 | 6
Chills (General disorders) | 6 | 1
Urinary tract infection (Infections and infestations) | 8 | 10
Upper respiratory tract infection (Infections and infestations) | 5 | 10
Sinusitis (Infections and infestations) | 10 | 4
Headache (Nervous system disorders) | 9 | 6
Multiple sclerosis relapse (Nervous system disorders) | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 2 | 6
Depression (Psychiatric disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.